CLINICAL TRIAL: NCT01201694
Title: Phase I Study of Surface-Controlled Water Soluble Curcumin (THERACURMIN CR-011L) in Patients With Advanced Malignancies
Brief Title: Phase I Study of Surface-Controlled Water Soluble Curcumin (THERACURMIN CR-011L)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other); Theravalues, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0276
Record Dates: First submitted 2010-09-09; First posted 2010-09-14 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Cancers
Keywords: Advanced malignancies; Surface-controlled water soluble curcumin; Turmeric; Dietary supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surface-Controlled Water Soluble Curcumin Group (Experimental): Starting dose 100 mg by mouth two times a day of a 28 day cycle.
  Interventions: Drug: Surface-Controlled Water Soluble Curcumin
- Surface-Controlled Water Soluble Curcumin Expansion (Experimental): Following finding of MTD surface-controlled water soluble curcumin, escalating dose levels
  Interventions: Drug: Surface-Controlled Water Soluble Curcumin MTD

INTERVENTIONS:
Drug: Surface-Controlled Water Soluble Curcumin — Starting dose 100 mg by mouth two times a day of a 28 day cycle.
  Arms: Surface-Controlled Water Soluble Curcumin Group
Drug: Surface-Controlled Water Soluble Curcumin MTD — Dose will be maximum tolerated dose (MTD) from Arm 1.
  Arms: Surface-Controlled Water Soluble Curcumin Expansion

SUMMARY:
The goal of this clinical research study is to find the highest tolerable doses of surface-controlled water dispersible curcumin (curcumin) that can be given to patients with advanced cancer. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Curcumin is the active ingredient in the spice, turmeric. It is a natural anti-inflammatory compound and has shown anti-tumor activity. Surface-controlled water dispersible curcumin is designed to be better absorbed by the body than regular curcumin.

Study Groups:

The first group of participants will receive the lowest dose level. Each new group will usually receive a higher dose than the group before it, if no intolerable side effects were seen. Each group will have 3-6 participants. This will continue until the highest tolerable dose of curcumin is found. Up to 6 dose levels of curcumin will be tested. Once the highest tolerable dose of each arm is found, up to 14 extra participants will be enrolled for extra safety testing.

In some cases, extra participants may be enrolled at dose levels shown to be safe for extra safety and/or pharmacokinetic (PK) and pharmacodynamic (PD) testing.

You will be assigned to a dose level based on when you join this study.

The dose of the study drug that you receive may be lowered if you have any intolerable side effects. If you are tolerating the treatment, your study drug dose may be increased after the first cycle to the highest dose level shown to be safe.

Study Drug Administration:

Each study "cycle" is 28 days long.

You will take 1 dose of curcumin on Day 1 of Cycle 1. Starting on Day 2 of Cycle 1, you will begin taking curcumin 2 times each day.

Curcumin is a liquid that comes in a bottle, and you will take it by mouth on an empty stomach with a full glass of water (8 ounces). If you are not tolerating the doses and your doctor thinks it is needed, you may take curcumin in divided doses several times a day with food.

Study Visits:

Before your first dose of study drug and during Week 2 of Cycle 2, you will complete a questionnaire about your quality of life. It should take about 5-10 minutes to complete.

Every week of Cycle 1 and then as often as the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for routine tests.

Before you begin each cycle:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any side effects you may be having.

At the end of Cycle 2 and then every 2-3 cycles:

* You will have a chest x-ray, CT, MRI, and/or PET scan to check the status of the disease. If the study doctor thinks it is needed, these scan may be performed more often. You also may have extra types of scans not listed in this consent form.
* If the doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.

PK Testing:

Blood (about ½ teaspoon each time) will be drawn for PK testing at the following times:

* On Day 1 of Cycle 1, blood will be drawn before the dose and then 6 more times over the next 6 hours after the dose.
* On Day 2 of Cycle 1, blood will be drawn 1 time.

Length of Study:

You may remain on study for as long as the study doctor thinks it is in your best interest. You will be taken off study early if the disease gets worse or you experience intolerable side effects.

Your participation on the study will be over once you have completed the end-of-study visit.

End-of-Study Visit:

Within 30 days after your last dose of the study drug(s), you will have an end-of-study visit. At this visit the following tests and procedures will be performed:

* Your medical history will be recorded.
* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* You will be asked about any side effects you may be having.
* If the study doctor thinks it is needed, you will have a chest x-ray, CT, MRI, and/or PET scan to check the status of the disease. If the study doctor thinks it is needed, you may also have extra types of scans.
* If the study doctor thinks it is needed, blood (about 1 teaspoon) will be drawn to measure tumor markers.

This is an investigational study. Curcumin is a commercially available substance, which is commonly used as a food additive. Curcumin is not FDA approved for any usage. At this time, curcumin is only being used in research.

Up to 72 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have an advanced malignancy that has either failed one or more prior therapies, or for which there is no established standard of care therapy that improves survival by at least 3 months. If standard therapies are available, the informed consent states that patients are forgoing approved therapies proven to prolong life or the time that the patient is alive without growth of their cancer.
2. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 3 or better (0-3).
3. Patients must have normal organ and marrow function as defined below: Absolute neutrophil count > 1,000 /uL Platelets > 50,000 /uL Total bilirubin </= 1.5 x upper limit of normal (ULN) (except patients with Gilbert's syndrome, who must have a total bilirubin < 3.0 mg/dL) and ALT </= 3 x ULN, Creatinine </= 1.5 x ULN or creatinine clearance >/= 40 ml/min
4. Patients must be able to understand and be willing to sign an Institutional Review Board (IRB) approved written informed consent document.
5. Women of child-bearing potential (women who are not postmenopausal for at least one year or are not surgically sterile) and men must agree to use adequate contraception (e.g., barrier device) prior to study entry, for the duration of study participation, and for 30 days after the last dose.
6. Patients may receive palliative radiation therapy immediately before or during the treatment if the radiation therapy is not delivered to the sole target lesions.
7. Men and women aged >/= 18 years. However, patients who are 13 years or older will be eligible after consultation with their pediatric attending.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure (NYHA Class III or IV), unstable angina pectoris, active bleeding that requires hospitalization, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Subject that has not recovered from major surgical procedure, open biopsy, or significant traumatic injury (i.e. subject still needs additional medical care for these issues).
3. History of gastric or duodenal ulcers, or hyperacidity syndromes.
4. History of allergic reactions to the study drug or its analogs.
5. Patient that has received any treatment for tumor specific control within 3 weeks of the start of study drug with investigational drugs and cytotoxic agents, or within 2 weeks of cytotoxic agent given weekly, or within 6 weeks of nitrosoureas or mitomycin C, or within 5 half-lives of biological targeted agents with half-lives and pharmacodynamic effects lasting less than 5 days (that includes, but is not limited to, erlotinib, sorafenib, sunitinib, bortezomib, and other similar agents).
6. Currently taking therapeutic doses of anticoagulants such as warfarin or antiplatelet agents (any prophylaxis agents are acceptable).
7. International normalized ratio (INR) > 1.5
8. Biliary obstruction or cholelithiasis.
9. Inability to take oral medication (PEG tube is acceptable).
10. Pregnant or breastfeeding women.
11. Concurrent enrollment on another therapeutic research study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Surface-Controlled Water Dispersible Curcumin | 4 weeks
  MTD defined by dose limiting toxicities (DLTs) that occur in the first cycle. DLT defined as treatment-related grade 3 or greater non-hematological toxicity other than nausea, vomiting, drug-related grade 3 or greater electrolyte abnormalities that do not return to ≤ grade 1 or baseline within 72 hours, or grade 3 nausea and vomiting related to study drug treatment that is not controlled at 72 hours despite appropriate antiemetic therapy. The defined events will be considered as DLT if they occur within the first cycle (28 days).

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org